CLINICAL TRIAL: NCT06278480
Title: Clinical Trial to Evaluate the Regeneration of Articular Cartilage Through Arthroscopy After MegaCarti® Application : Multicenter, Comparative, Evaluator-blinded, Retrospective Study
Brief Title: Clinical Trial to Evaluate the Regeneration of Articular Cartilage Through Arthroscopy After MegaCarti® Application
Status: Completed | Type: Observational
Sponsor: L&C Bio (Industry)
Responsible Party: Sponsor
Other Study IDs: LNC-MECA-003
Record Dates: First submitted 2024-01-25; First posted 2024-02-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MegaCarti®: Experimental: MegaCarti® application after microfracture The experimental group is applied with MegaCarti® and underwent high tibial osteotomy(HTO) after microfracture.
  Interventions: Device: MegaCarti®; Procedure: microfracture
- Microfracture only: The control group underwent microfracture and high tibial osteotomy(HTO)
  Interventions: Procedure: microfracture

INTERVENTIONS:
Device: MegaCarti® — Medical devices containing allogeneic cartilage
  Groups: MegaCarti®
Procedure: microfracture — microfracture

SUMMARY:
The MegaCarti® is the decellularized allogeneic cartilage and acts as a cover after bone marrow stimulation to prevent the loss of blood clots and induces cartilage regeneration by assisting in the location of stem cells derived from bone marrow. During the 48-week confirmatory clinical trial of MegaCarti®, patients who simultaneously underwent high tibial osteotomy(HTO) were treated with a group in which MegaCarti® was implanted after microfracture and a group in which microfracture alone was performed. Cartilage regeneration is evaluated in patients with arthroscopy data at the time of fixation removal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients participating in the "Clinical Trial to Evaluate the Efficacy and Safety of MegaCarti® ; Cartilage Defect Treatment Assisting Cartilage Regeneration in Knee Cartilage Defects : Multicenter, Independent Evaluator and Subject Blinded, Microfracture Comparative, Superiority, Randomized, Confirmatory Clinical Study and 5 Years Follow up Study"
2. Patients who simultaneously underwent HTO during knee joint cartilage surgery

Exclusion Criteria:

N/A

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The MegaCarti® is the decellularized allogeneic cartilage and acts as a cover after bone marrow stimulation to prevent the loss of blood clots and induces cartilage regeneration by assisting in the location of stem cells derived from bone marrow. During the 48-week confirmatory clinical trial of MegaCarti®, patients who simultaneously underwent HTO were treated with a group in which MegaCarti® was implanted after microfracture and a group in which microfracture alone was performed. Cartilage regeneration is evaluated in patients with arthroscopy data at the time of fixation removal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Comparison of the ICRS-Cartilage Repair Assessment grade-Overall repair assessment | When removing fixtures after HTO (an average of 1 year after surgery)
  Primary Endpoint [experimental group / control group]
Comparison of macroscopic status of regenerated cartilage | When removing fixtures after HTO (an average of 1 year after surgery)
  Primary Endpoint [experimental group / control group]

SECONDARY OUTCOMES:
Comparison of IKDC score | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group], Higher scores mean a better outcome
Comparison of VAS score | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group], Higher scores mean a worse outcome
Comparison of KOOS score | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group], Higher scores mean a better outcome
Comparison of WOMAC score | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group], Higher scores mean a worse outcome
Comparison of Kellgren-Lawrence grade | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group]
Comparison of HKA angle, Posterior Tibial slope | At last visit (an average of two years after surgery)
  Secondary Endpoint [experimental group / control group]

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Gangnam Severance Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No